CLINICAL TRIAL: NCT05157776
Title: Neoadjuvant Sintilimab and Platinum-based Chemotherapy for Resectable Locally Advanced NSCLC Harboring no Driver Mutations: A Prospective, Randomized, Multicenter Phase III Trial
Brief Title: A Phase III Trial of Neoadjuvant Sintilimab and Chemotherapy for NSCLC Harboring No Driver Mutations
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Jiang Fan, Director of Department of Thoracic Surgery, Tongji University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGHDOT 21-10
Record Dates: First submitted 2021-12-07; First posted 2021-12-15 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: NSCLC, Stage IIIA; EGF-R Negative Non-Small Cell Lung Cancer; ALK Negative NSCLC
Keywords: Neoadjuvant; PD-1; NSCLC; Phase III; Platinum-based; Locally Advanced
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Neoadjuvant therapy of Sintilimab and chemotherapy in 2 cycles before surgery and optional adjuvant therapy of Sintilimab and chemotherapy in 2 cycles after surgery
  Interventions: Drug: PD-1 and chemotherapy
- Experimental group (Experimental): Neoadjuvant therapy of Sintilimab and chemotherapy in 4 cycles before surgery
  Interventions: Drug: PD-1 and chemotherapy

INTERVENTIONS:
Drug: PD-1 and chemotherapy — Sintilimab+(Squamous)ABX+DDP/CBP, or (non-Squamous)PEM+DDP/CBP

SUMMARY:
This is a randomized, open-label study designed to evaluate the safety and efficacy of neoadjuvant PD-1 antibody plus chemotherapy followed by surgery in resectable stage IIIA non-small cell lung cancer.

The primary endpoint: pCR rate The second endpoint: MPR, DFS, MRD

DETAILED DESCRIPTION:
This study is a prospective, multicenter, phase III randomized controlled clinical study. Stage IIIA NSCLC patients with EGFR mutation negative and ALK rearrangement negative were enrolled, and after 2 courses of treatment with Sintilimab combined with Platinum-based Chemotherapy, they were randomly assigned 1:1 to the control group (surgical resection and postoperative treatment for 2 courses are recommended) or the experimental group (surgery after 2 courses of treatment).

The primary endpoint is pCR rate. The second endpoints are MPR, DFS, and MRD.

ELIGIBILITY:
Inclusion Criteria:

1. Resectable stage IIIA NSCLC, EGFR mutation-negative and ALK rearrangement negative (8th UICC TNM staging);
2. No prior anti-tumor therapy for NSCLC;
3. Age from 18 to 75 years old;
4. Adequate organ function:

   Hemoglobin ≥9.0g/L; White blood cell count 4.0~10×109/L; The absolute value of neutrophils (ANC) ≥ 1.5×109/L; Platelet count ≥100×109/L; Total bilirubin ≤ 1.5 times the upper limit of normal; ALT and AST≤2.5 times the upper limit of normal; The international normalized ratio of prothrombin time is ≤1.5 times the upper limit of normal value, and the partial thromboplastin time is within the range of normal value; Creatinine ≤ 1.5 times the upper limit of normal;
5. No chemotherapy, radiotherapy or hormone therapy for malignant tumors, no history of other malignant tumors, excluding patients who have received hormone therapy for prostate cancer and have had DFS for more than 5 years;
6. ECOG 0～1;

Exclusion Criteria:

1. Double primary or multiple primary NSCLC;
2. EGFR mutation or ALK mutation was positive
3. patients with psychosis;
4. Pre-existing or coexisting bleeding disorders;
5. Other uncontrollable and inoperable patients;
6. Patients whose previous operations have prevented this operation from being performed;
7. Female patients who are pregnant or breastfeeding;
8. For patients who are allergic to the drugs in the program.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Pathologically complete response (pCR) rate | in three weeks after the surgical resection

SECONDARY OUTCOMES:
Major pathological response (MPR) rate | in three weeks after the surgical resection
Disease-free survival (DFS) | one, two, three and five years since the initial treatment (each treatment is 2 days)
Minimal residual disease(MRD) | in one week before each cycle and in the forth week after the surgical resection (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Fan, MD, Principal Investigator — Shanghai General Hospital; Shanghai Pulmonary Hospital
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin D, Wu L, Wang P, Li X, Wang X, Cai Y, Xiong K, Chen X, Yang F, Huang W, Wang X, Fan J. Dynamic circulating tumor DNA indicates pathological benefits of additional neoadjuvant chemoimmunotherapy courses for locally advanced non-small-cell lung cancer patients. Front Oncol. 2025 Jul 24;15:1563315. doi: 10.3389/fonc.2025.1563315. eCollection 2025. PMID 40777124